CLINICAL TRIAL: NCT02513914
Title: Operative Procedures Vs. Endovascular Neurosurgery for Untreated Pseudotumor Trial (OPEN-UP)
Brief Title: Operative Procedures Vs. Endovascular Neurosurgery for Untreated Pseudotumor Trial
Acronym: OPEN-UP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has suspended the study and is not enrolling any new participants. It is due to funding unavailability.
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Barrow Neurological Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15BN045
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2024-05

CONDITIONS: Pseudotumor Cerebri; Idiopathic Intracranial Hypertension (IIH)
Keywords: endovascular neurosurgery
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dural Venous Sinus Stenting (Experimental): Pt. will undergo pre-treatment with aspirin and clopidogrel. Transfemoral venous access will be obtained (pt. heparinized).Guide catheter will be placed in jugular bulb ipsilateral to dural venous sinus stenosis. Stent will be deployed across stenotic segment. Balloon angioplasty will not be performed unless initial stenosis is not easily traversed with stent. No pressure measurements will be taken during stent placement. Patients will undergo serial physical/neuro exams for 24 hours post-procedure. Daily dual anti-platelet treatment will continue for 6 months after initial procedure, after which clopidogrel will be discontinued and aspirin 81mg daily will be prescribed indefinitely. If significant bilateral venous sinus stenosis is present, stenosis with more severe pressure gradient will be stented. In pt. with bilateral venous sinus stenosis with equivalent pressure gradients, side will be at surgeon's discretion.
  Interventions: Device: Dural Venous Sinus Stenting
- Cerebrospinal Fluid Shunting (Active Comparator): Choice of shunt procedure (ventriculoperitoneal, ventriculoatrial, or lumboperitoneal), catheter laterality, brand and shunt equipment (including shunt catheters and valves), valve settings of programmable shunt valves (when applicable), intrathecal antibiotic administration and the use of stereotactic navigation will be at the discretion of neurosurgeon. Shunt procedures will be performed per the standard of care, under general anesthesia. An optional surgical procedure guidance document will be provided for other sites. Patients will undergo serial physical and neurological examinations for 24 hours post-procedure prior to discharge.
  Interventions: Device: Cerebrospinal Fluid Shunting

INTERVENTIONS:
Device: Dural Venous Sinus Stenting — See Dural Venous Sinus Stenting arm.
  Arms: Dural Venous Sinus Stenting
Device: Cerebrospinal Fluid Shunting — See Cerebrospinal Fluid Shunting arm.
  Arms: Cerebrospinal Fluid Shunting

SUMMARY:
Pseudotumor cerebri, also called idiopathic intracranial hypertension (IIH), is characterized by elevated intracranial pressure, headache, and if severe, vision loss. IIH is difficult to treat. Medical management may not adequately resolve the symptoms, and surgical management (primarily through cerebrospinal fluid [CSF] shunting) has a high failure rate. Recently, a relationship between IIH and stenosis of the dural venous sinuses (the veins that drain blood from the brain) has been reported. In patients with IIH in whom there is stenosis of one or more dural venous sinuses, placing a stent in the venous sinus may improve patients' objective symptoms (such as visual loss and papilledema) and subjective symptoms (such as headache). This study will determine whether dural venous sinus stenting is as effective as CSF shunting (considered the standard surgical treatment) in treating IIH patients who have moderate vision loss and stenosis of the dural venous sinuses.

DETAILED DESCRIPTION:
Screening evaluation: Screening will include standard-of-care IIH evaluation including general medical and neurological examinations, blood chemistries, complete blood count, prothrombin time (PT),partial thromboplastin time (PTT), and pregnancy test. Ophthalmological evaluation will include visual acuity, pellucid marginal degeneration (PMD), and optical coherence tomography (OCT). Quality of life assessments are Headache Impact Test-6, Short Form Health Survey-36 and Visual Function Questionnaire-25 + Neuro-Ophthalmology supplement tests. Participants must have had a recent (within 6 months of enrollment) magnetic resonance imaging (MRI) of the brain as well as a diagnostic lumbar puncture (including opening pressure, cerebrospinal fluid (CSF) cell count, CSF glucose and CSF protein), both of which are also part of the standard of care for diagnosis of IIH.

Eligible patients will undergo outpatient diagnostic venography within one month of initial IIH evaluation. Under local anesthesia, transfemoral venous access will be obtained and a guide catheter will be placed in the right jugular bulb. A microcatheter (Excelsior SL-10, Stryker Neurovascular) will then be advanced into the dural venous sinuses, and venography will be performed to determine the presence of any dural venous sinus stenosis. Then, blood pressure will be transduced through the microcatheter at the following anatomic locations: Anterior superior sagittal sinus, posterior superior sagittal sinus, bilateral transverse sinuses, bilateral sigmoid sinuses and bilateral jugular bulbs. The venous pressure gradient will be defined as the difference in pressure measurements between the anatomic locations proximal and distal to any stenotic venous sinus segment, or between the transverse and sigmoid sinuses. A pressure gradient of ≥ 8 mmHg is considered sufficient for subsequent randomization. In patients in which pressure gradient is < 8 mmHg, the patient will not be randomized.

Subsequent visits: Once a patient has met eligibility criteria and undergone randomization, treatment will occur within one month of the Neuro-Ophthalmology evaluations and within one month of diagnostic venography. Follow-up visits will occur at post procedure prior to discharge (24 hours), two weeks, six months and one year after the index procedure.

At post-procedure follow-up, patients will undergo physical and neurological exams. At two-week follow-up (within one week on either side), patients will undergo neurological and ophthalmological evaluations, OCT, perimetry, and visual acuity testing for safety. While perimetry at this point will not be used for primary outcome analysis, substantial worsening in any of the above measures despite treatment will prompt consideration for treatment failure.

At six-month follow-up, subjects will undergo perimetry for primary outcome analysis, outpatient diagnostic cerebral venography, and pressure measurements identical to that of the screening evaluation (including pressure measurements at all predefined anatomical locations) within four weeks on either side of the six-month target date. At both six-month and one-year follow-up visits, patients will complete follow-up quality of life questionnaires (HIT-6, SF-36 and VFQ-25 + Neuro-Ophthalmology supplement).These visits will also include queries regarding interim medical history, headache status, medication usage (specifically details and dose of those agents used to treat IIH or headache), and the number of IIH-related procedures each subject has undergone since the index procedure. At one-year follow-up, the patient will undergo Magnetic Resonance Venography (MRV) or Computed Tomography Venography (CRV) to assess patency of stented dural sinus. Follow-up will occur within four weeks on either side of the one-year target date.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Diagnosis of Idiopathic Intracranial Hypertension according to the Modified Dandy Criteria.
* Moderate to severe visual field loss defined by perimetric mean deviation of at least -8 dB but better than -30 dB in the worst eye.
* Diagnostic cerebral venography demonstrating a pressure gradient of ≥ 8 mmHg across at least one segment of the dural venous sinus as measured during transfemoral cerebral venography
* Failure of conservative or non-surgical therapies,by:

  1. failed medical treatment including weight loss regimens OR
  2. medication intolerance OR
  3. medical treatment not indicated per investigator team
* Women must not be able to become pregnant (e.g., post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study, and have a negative pregnancy test prior to treatment.

  a. Women on hormonal birth control must be on a stable dose for at least 3 months prior to enrollment
* Signed informed consent obtained from the patient.

Exclusion Criteria:

* CSF pressure <25 cm H2O on lumbar puncture.
* Abnormal CSF analysis such as elevated protein (>60 mg/dL), low glucose (<30 mg/dL), elevated cell count >5 (unless traumatic lumbar puncture).
* Previous CSF shunt or diversion procedure of any kind, or previous optic nerve sheath fenestration.
* Uncontrolled second primary headache disorder (e.g. chronic migraine, medication overuse headache).
* Allergic reaction to radiological iodine contrast agent.
* Significant renal impairment (serum creatinine >1.5 mg/dL).
* Contraindication to general anesthesia.
* Contraindication to aspirin, clopidogrel or other anticoagulants.
* Presence of a cranial vascular abnormality (arteriovenous malformation, dural arteriovenous fistula, dural venous sinus thrombosis) or other intracranial mass.
* Presence of a hypercoagulable state such as Factor V Leiden, Protein C or S deficiency or anti-cardiolipin syndrome.
* Inability to provide reliable and reproducible visual field examinations (>15% false- positive errors and/or failure to maintain fixation for eye monitoring).
* Previous or ongoing eye disease such as glaucoma or retinopathy.
* Pre-existing best corrected visual acuity worse than 20/200 in the study eye as measured by Snellen charts, without meeting eligible ophthalmological criteria in the contralateral eye.
* Other pre-existing conditions accounting for optic atrophy that could produce irreversible vision loss in the study eye without meeting eligible ophthalmological criteria for IIH in the contralateral eye.
* Condition associated with high risk of retinopathy (e.g. type I diabetes).
* Previously (within the last 2 months) or currently exposed to a drug or substance that may elevate intracranial pressure (e.g. lithium, high-dose vitamin A, tetracyclines, anabolic steroids, chlordecone, amiodarone, diphenylhydantoin, nalidixic acid).
* Pregnancy.
* Presence of a physical, mental or social condition that could prevent adequate follow-up such as terminal illness, homelessness, lack of telephone, drug dependency or anticipation of a significant move away from a study site within one year of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Perimetric mean deviation (PMD) at six months | Six months
  PMD was chosen as a primary outcome due to its generalizability, test-retest reliability and standardization across centers, as well as its sensitivity to severity and progression of visual symptoms of IIH. Based on previous work by the Neuro-Ophthalmology Research Disease Investigator Consortium (NORDIC) investigators, we defined the upper and lower bounds of visual field loss severity for study inclusion as between -8 and -30 dB in the worst-affected eye. The upper limit of -8 dB ensures enough baseline visual loss to consider surgical treatment and allow room for improvement, while the lower limit of -30 dB ensures that patients with severe visual loss unlikely to significantly improve with any treatment would be excluded. PMD will be tested using Swedish Interactive Threshold Algorithm (SITA) standard 24-2 perimetry with stimulus size III.

SECONDARY OUTCOMES:
Total number of IIH-related surgeries at one year | Six months and One year
  The number of revision surgeries includes either additional stenting for any reason in the stent group, shunt revision for any reason in the shunt group, or other IIH procedures such as optic nerve sheath fenestration in either group. The total number of procedures will be assessed at one year from the index procedure.
Papilledema | Study entry, two-weeks post-operative and six months
  Papilledema will be measured by OCT, as it is considered more quantitative than fundus photography or Frisén grading.
Quality of life | Study entry, six months and One year
  Both headache and visual quality of life instruments will be used to assess subjective measures of treatment impact. These include the HIT-6 headache and SF-36 scales for disability assessment, as well as the VFQ-25 questionnaire (plus the 10 question Neuro-Ophthalmology supplement) for visual disability.
Medication usage | Two-weeks post-operative, six months and One year
  A simple binary choice of reduced or unchanged/increased usage of headache-modifying medications (including narcotic and non-narcotic analgesics and muscle relaxants)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe C Albuquerque, MD, Principal Investigator — Barrow Neurosurgical Associates
Locations (2):
- United States (2):
  - Barrow Neurological Institute at Dignity Health St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - University of Washington Department of Neurosurgery, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No